CLINICAL TRIAL: NCT03281564
Title: Prospective Study of Quality of Life After Laparoscopic Removal of Essure®
Brief Title: Quality of Life After Laparoscopic Removal of Essure®
Acronym: ABLIMCO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0479
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-05

CONDITIONS: Contraceptive Device; Complications; Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Essure®: Patients with laparoscopic removal of Essure®
  Interventions: Other: Quality of life after Essure® removal

INTERVENTIONS:
Other: Quality of life after Essure® removal — Questionnaire to assess the quality of life 1, 3, 6 and 12 months after laparoscopic removal of Essure® device

SUMMARY:
A lot of patients seem to complain after hysteroscopic tubal occlusion by Essure® device with a worce quality of life. Investigators' hypothesis is that Essure® laparoscopic removal may improve quality of life. This prospectice study aim to assess the quality of life 1, 3, 6 and 12 months after Essure® removal.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18 years or more
* patients with Essure® sterilization device
* surgical removal of Essure® with bilateral salpingectomy by laparoscopy

Exclusion Criteria:

* interview revealing disorder entailing unacceptable risk of postoperative complications: coagulation disorder, immune system disorder, evolutive disease, etc.
* impaired lower-limb range of motion preventing positioning for surgery
* inability to understand information provided
* prisoner or under administrative supervision.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with laparoscopic removal of Essure®
Sampling Method: Non-Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2017-10-14 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Quality of life 1 month after laparoscopic removal of Essure® | 1 month
  Questionnaire to assess the quality of life 1 month after laparoscopic removal of Essure® device

CONTACTS AND LOCATIONS:
Locations (1):
- Gynaecology Department, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trecourt A, Devouassoux-Shisheboran M, Nohuz E, Cerruto E, Moret S, Hallez D, Miguet-Bensouda C, Chene G. Clinical and histopathological correlations in symptomatic patients with salpingectomy for Essure(R) implant removal: a cross-sectional study. Eur J Contracept Reprod Health Care. 2023 Aug;28(4):227-233. doi: 10.1080/13625187.2023.2218953. Epub 2023 Jun 27. PMID 37365993